CLINICAL TRIAL: NCT03424057
Title: A Novel Technique in the Treatment of Sacrococcygeal Pilonidal Sinus Disease: Effect of Reduction of Dead-space With Asymmetric Primary Closure and Additional Skin Excision Technique.
Brief Title: Asymmetric Primary Closure and Additional Skin Excision Technique.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siverek Devlet Hastanesi (Other)
Responsible Party: Principal Investigator, Abdulcabbar Kartal, General surgeon, Siverek Devlet Hastanesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 74059997.050.01.04/79
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Pilonidal Sinus; Pilonidal Disease of Natal Cleft; Surgical Technique
Keywords: Karydakis modification; pilonidal sinus; seroma
MeSH Terms: conditions — Pilonidal Sinus; Seroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 were treated with the new technique (Asymmetric Primary Closure and Additional Skin Excision).
  In this new technique, following total sinus excision, the excision defect was closed with the standard Karydakis method, but an advancement tissue flap was performed using additional skin excision, in order to reduce the dead-space volume.
  Interventions: Procedure: Asymmetric Primary Closure and Additional Skin Excision Technique
- Group 2 (Active Comparator): Group 2 were treated with the standard Karydakis technique.
  Interventions: Procedure: Standard Karydakis technique.

INTERVENTIONS:
Procedure: Asymmetric Primary Closure and Additional Skin Excision Technique — In this new technique, following total sinus excision, the excision defect was closed with the standard Karydakis method, but an advancement tissue flap was performed using additional skin excision, in order to reduce the dead-space volume.
  Arms: Group 1
Procedure: Standard Karydakis technique. — In this new technique, following total sinus excision, the excision defect was closed with the standard Karydakis method
  Arms: Group 2

SUMMARY:
The aim of this study was to reduce the residual dead-space volume with a modification following the standard Karydakis procedure.

DETAILED DESCRIPTION:
All patients were operated in the jack-knife position under spinal anesthesia (SA). The gluteal parts of the patients were stretched in both directions with bandage and intergluteal cleft was opened. Methylen blue was administered from the sinus openings in the gluteal region. Then, total sinus excision was performed, including the entire sinus tracts by passing the skin, subcutaneous tissues up to the presacral fascia.

In patients operated with standard Karydakis procedure, a flap (Karydakis flap) extending along the incision was prepared, with the medial side of the wound to be 1 cm deep and 2-3 cm inward. The prepared flap was shifted to medial and sutured to the presacral fascia with 2/0 vicryl.

In patients who were operated with the Asymmetric Primary Closure with Skin Excision Technique, after the Karydakis flap was formed, 5-10 mm skin was excised along the incision from the side of the flap to reduce the volume of the dead-space laterally.

In both groups, subcutaneous tissue was approximated with 2/0 vicryl. The skin was sutured with mattress technique using 2/0 Prolene. No drains were used in patients from either group.

Patients were followed up for wound leakage, seroma and hematoma formation, skin dehiscence and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* All patients between age of 18-65 who had chronic pilonidal disease

Exclusion Criteria:

* Patients who did not accept the procedure
* Patients had undergone previous pilonidal sinus surgery
* Patientshad active infection
* Patients who were not minimum of 18 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2016-03-25 (Actual); Study Completion 2016-04-15 (Actual)

PRIMARY OUTCOMES:
Early postoperative complications. | 3 years
  wound dehiscence, formation of seroma, hematoma, wound infection

IPD SHARING:
Plan to Share IPD: Yes
The study has been completed. The datas will be shared as an article
Supporting Information: Study Protocol, SAP, CSR